CLINICAL TRIAL: NCT06540001
Title: Development and Validation of an Automated Self-administered Visual Acuity System
Acronym: AutoVA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Singapore Institute of Technology (Other); Nanyang Technological University (Other); Lee Kong Chian School of Medicine, Nanyang Technological University (Unknown)
Responsible Party: Principal Investigator, Li Zhenghao Kelvin, Consultant, Tan Tock Seng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024/00157
Record Dates: First submitted 2024-07-27; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Visual Impairment
Keywords: Visual acuity
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will undergo both automated and manual visual acuity testing (Experimental): Patient will perform manual visual acuity first, then be guided to another room to have the visual acuity tested on the automated VA device
  Interventions: Device: Automated visual acuity

INTERVENTIONS:
Device: Automated visual acuity — The automated visual acuity device is developed in collaboration with Tan Tock Seng Hospital, Singapore Institute of Technology and Nanyang Technological University. It uses artificial intelligence for pose estimation and speech recognition to infer if the participant is reading the correct letters displayed on the screen.

SUMMARY:
Visual acuity tests, commonly conducted in clinics and used for health screenings, are becoming more in demand due to an aging population. Current online self-eye check apps are limited as they don't accurately reflect true distance vision assessed in clinical settings. These tests, performed by trained personnel, are time-consuming and can cause delays in clinics. This project aims to develop an automated Visual Acuity (VA) station using AI technologies like speech-to-text and computer vision, hypothesizing that it can match the accuracy of manual assessments by clinic staff, thus potentially reducing waiting times and improving efficiency.

DETAILED DESCRIPTION:
Visual acuity is done as a routine eye check for the majority of eye patients in the clinic. It is also done as a screening test for pre-employment health checks and health screening. Patients can be checked for refractive errors, on a community level or screened for eye diseases, for those with chronic medical conditions. With the increasing burden of aging population and eye conditions, the number of patients in eye clinics will increase.

There are a few existing online applications that allow self-eye checks, however there are limitations. They are usually done at an intermediate distance, i.e. distance from phone to eye and does not accurately represent true distance vision. Distance vision is typically set at 4- 6m in a clinical setting.

A visual acuity test is administered by specially trained healthcare personnel, such as optometrists and patient service assistants, which is often time-consuming and labour intensive, where one-on-one attention is required. In addition, vision is subjective and re-testing may be required at times to ensure accurate vision assessment.

As the visual acuity test is the first clinical station patient goes to after registration, this leads to a bottleneck in workflow causes delays in the subsequent services and eventually increases patient waiting times in the clinics.

This project aims to develop and validate an automated Visual Acuity (VA) station through speech-to-text and computer vision technology in comparison to existing manual VA assessments.

We hypothesize that we are able to use artificial intelligence to understand patient's speech and posture to automate the visual acuity test. We also hypothesize that the automated visual acuity test is comparable to having VA checked manually by a clinic staff.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age >21 and able to give consent
2. Patients who have at least counting finger vision
3. Patients who is able to speak in an audible and clear voice
4. Patients who is able to use a digital device independently (e.g. handphone)

Exclusion Criteria:

1. Patients on wheelchair/ walking aids
2. Patients with hearing difficulties
3. Patients with speech difficulties
4. Patients who have cognitive impairment
5. Patients who are hemiplegic/ motor dysfunction
6. Patients who have vision worse than counting fingers
7. Patients who are pregnant

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity with and without pinhole using Snellen letters and numbers | 1 year
  Best corrected visual acuity will be expressed in metres (e.g. 6/6-1), and will be converted to LogMAR for analysis.

IPD SHARING:
Plan to Share IPD: No